CLINICAL TRIAL: NCT04939116
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of Safety and Efficacy of ANG-3070 in Patients With Primary Glomerular Disease and Persistent Proteinuria
Brief Title: Study of Safety and Efficacy of ANG-3070 in Chronic Kidney Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Angion Biomedica Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANG3070-CKD-201
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Glomerular Disease; Proteinuria
Keywords: Glomerular Disease; Chronic Kidney Disease; Proteinuria
MeSH Terms: conditions — Proteinuria; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 200 mg QD (Experimental): 200 mg of ANG-3070 will be taken once daily for 12 weeks.
  Interventions: Drug: ANG-3070
- 400 mg QD (Experimental): 400 mg of ANG-3070 will be taken once daily for 12 weeks
  Interventions: Drug: ANG-3070
- 300 mg BID (Experimental): 300 mg of ANG-3070 will be taken twice a day for 12 weeks.
  Interventions: Drug: ANG-3070
- Placebo (Placebo Comparator): Placebo capsules will be taken once or twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANG-3070 — Orally administered tyrosine kinase inhibitor capsule
  Arms: 200 mg QD; 300 mg BID; 400 mg QD
Drug: Placebo — Orally administered placebo capsule
  Arms: Placebo

SUMMARY:
The major objective is to demonstrate the safety and efficacy of ANG-3070 in patients with primary glomerular disease and persistent proteinuria.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of ANG-3070 in patients with primary glomerular disease and persistent proteinuria while on the SOC, as measured by a reduction in the 24-hour urinary protein excretion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 and older.
2. Diagnosis of a primary glomerular disease confirmed from a past renal biopsy. Participants with genetic forms of FSGS may be enrolled without a renal biopsy if the clinical picture is consistent with the genetic testing results.
3. Estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) ≥ 40 mL/min/1.73m2.
4. Urinary protein excretion ≥ 1 g/day on a 24-hour urine collection.
5. All participants must be on the SOC therapy, including the maximally tolerated/recommended doses of an ACEi or ARB, but not both.

Exclusion Criteria:

1. Positive Hepatitis B (HBV), Hepatitis C (HCV), or human immunodeficiency virus (HIV) viral screening; historical or during screening.
2. Aspartate Aminotransferase (AST) or alanine Aminotransferase (ALT) or total bilirubin > 2 x ULN.
3. Hemoglobin A1C > 8.5%.
4. Known predisposition to bleeding and/or thrombosis
5. Type I diabetes mellitus.
6. Renal disease secondary to systemic disease including but not limited to: systemic lupus erythematosus, anti-neutrophil cytoplasmic antibodies -associated diseases, anti-glomerular basement disease, secondary forms of focal segmental glomerulosclerosis, renal diseases associated with para-proteinemias, C3 glomerulopathy, and diabetic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in 24-hour urinary protein excretion at Week 12 | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: John Neylan, MD, Study Director — Angion Biomedica
Locations (29):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Amicis Reserach Center, Northridge, California
  - Amicis Reserach Center, Vacaville, California
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Genesis Clinical Research LLC, Tampa, Florida
  - Davita Clinical Research, Columbus, Georgia
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Davita Clinical Research, Edina, Minnesota
  - Clinical Research Consultants, LLC., Kansas City, Missouri
  - Frenova Renal Research/Nephrology and Hypertension Specialists, St Louis, Missouri
  - St. Louis Kidney Care, St Louis, Missouri
  - New Jersey Kidney Care, Jersey City, New Jersey
  - NYU Langone Nephrology Associates, Mineola, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Prolato Clinical Research Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- Australia (6):
  - Nepean Hospital, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Melbourne, Victoria
  - Western Hospital, Saint Albans, Victoria
- Georgia (5):
  - JSC "Evex Hospitals", Kutaisi
  - LtD Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - "Tbilisi State Medical University's and Ingorokva's University Clinic of High Medical Technologies" LTD, Tbilisi
  - Ivane Bokeria Tbilisi Referral Hospital, Tbilisi
  - Tbilisi Heart Center, Tbilisi